CLINICAL TRIAL: NCT05784467
Title: Addressing Intersectional Stigma Through Coping, Resistance, and Resilience to Improve Methamphetamine Use and Factors Influencing PrEP Uptake Among Latino MSM: a Step Towards Ending HIV by 2030
Brief Title: Methamphetamine, PrEP, and Intersectional Stigma Study
Acronym: eMPrISe
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1K01DA055521 (NIH)
Record Dates: First submitted 2023-03-13; First posted 2023-03-27 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Methamphetamine Abuse; Hiv; Social Stigma
Keywords: Methamphetamine; Preexposure prophylaxis; Intersectional Stigma
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Social Stigma | interventions — Methamphetamine

STUDY DESIGN:
Intervention Model Description: Each group will receive the same intervention components, but one group will be facilitated in English and the other, Spanish.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- English (Other): Participants in the English arm will receive the eMPrISe intervention materials in English.
  Interventions: Behavioral: Methamphetamine, PrEP, and Intersectional Stigma (eMPrISe) study
- Spanish (Other): Participants in the English arm will receive the eMPrISe intervention materials in Spanish.
  Interventions: Behavioral: Methamphetamine, PrEP, and Intersectional Stigma (eMPrISe) study

INTERVENTIONS:
Behavioral: Methamphetamine, PrEP, and Intersectional Stigma (eMPrISe) study — Group behavioral intervention with 12 weekly sessions lasting 2 hours focusing on coping, resistance, and resilience.

SUMMARY:
The goal of this clinical trail is to test the developed eMPrISe study in HIV-negative, adult, Latino men who have sex with men (MSM) who use non-injection substances. The main questions it aims to answer are:

* Can participation in the developed eMPrISe study reduce methamphetamine ('meth') use risk?
* Can participation in the developed eMPrISe study improve preexposure prophylaxis (PrEP) cascade progression? Participants will participate in 12 weekly modules that: (1) build critical thinking skills, (2) identify and discuss the link between oppression and harmful behaviors, (3) take action, (4) voice and validate feelings and experiences, and (5) share knowledge and resources.

DETAILED DESCRIPTION:
This is a clinical trial research experience to support Dr. Angel B Algarin's training. Findings from secondary analyses from AIMs 1 & 2 will guide the selection and adaptation of evidence-based, multi-level coping resistance and resilience intervention strategies to reduce the harmful effects of intersectional stigma on meth use and PrEP cascade progression.

Resistance: I plan to adapt Community Wise which is a 12-week multi-level, group intervention that moves participants from a cycle of oppression, feelings of powerlessness, and health risk behaviors to a cycle of empowerment, self-efficacy, and health promoting behaviors. The intervention was found to be effective in reducing recent substance use.

Coping: I plan to integrate effective components of the Effective Skills to Empower Effective Men (ESTEEM) study which utilizes a cognitive based therapy (CBT) approach to enhance stigma coping among MSM and has been found effective in reducing drug use and sexual risk behaviors.

Resilience: I plan to integrate resilience intervention strategies from the HealthMpowerment study which is grounded in the Institute of Medicine's Integrated Model of Behavior Theory and has been shown to reduce sexual risk behaviors and stigma among MSM.

The eMPrISe study will be developed using the ADAPT-ITT (Assessment, Decision, Adaptation, Production, Topical experts, Integration, Training, Testing) model and will be formatively evaluated among n=20 Latino MSM (10 English speaking & 10 Spanish speaking) with moderate meth use risk scores determined by Alcohol, Smoking and Substance Involvement Screening Test (ASSIST). Quantitative data will be collected via Qualtrics and Network Canvas for a 60-minute interviewer driven survey pre- and post-evaluation of adapted intervention, and for 10-minute self-administered questionnaires following each of the 12 modules. Qualitative data will be collected via audio recordings of participants' real time responses as they progress through the intervention to assess feasibility of the 12 weekly modules. Quantitative results will also inform semi-structured focus groups (1 English, 1 Spanish) to contextualize the acceptability of each of the 12 intervention modules and the intervention as a whole. While the formative evaluation will assess trends, it is not powered to detect pre-post changes in these measures.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* cisgender male
* self-identify as Latino or Hispanic
* fluent in English or Spanish
* any sexual activity with men in the past 12 months
* HIV-negative
* moderate methamphetamine use risk (as determined by the the ASSIST assessment)
* experience of intersectional stigma within their social network in the past 12 months
* willing to provide written informed consent

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender men
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Methamphetamine use risk | 3 Months
  Assessed using the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) Scores range from 0 - 39, where higher scores indicate higher risk.
PrEP cascade progression | 3 Months
  Assessed using the Motivational PrEP Cascade Ordinal outcome including: 1= PrEP pre-contemplation, 2= PrEP contemplation, 3=PrEParation, 4=PrEP Action & Initiation, 5=PrEP Maintenance

SECONDARY OUTCOMES:
Resistance | 3 Month
  Assessed using items adapted from the Stigma Resistance Scale Scores range from 0 - 76, where higher scores indicate higher levels of resistance
Resilience | 3 Month
  Assessed using items from the Connor-Davidson Resilience Scale (CD-RISC) Scores range from 0-40, where higher scores indicate higher levels of resilience
Coping | 3 Month
  Assessed using the Coping Inventory for Stressful Situations (CISS) Scores range from 0-84, where higher scores indicate higher levels of coping

IPD SHARING:
Plan to Share IPD: No